CLINICAL TRIAL: NCT01190228
Title: Assessment of the Memory Immune Response, Safety of Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Children Previously Immunized With a Single Dose of JE-CV and Long-Term Follow-Up
Brief Title: Study of Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Children Previously Immunized With JE-CV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEC15; UTN: U1111-1113-3629 (Other: WHO)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Japanese Encephalitis; Varicella
Keywords: Japanese Encephalitis; Japanese encephalitis chimeric virus vaccine; Varicella; Varicella vaccine
MeSH Terms: conditions — Encephalitis, Japanese; Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Intervention Model Description: This was an open, controlled, multicenter, Phase III trial. Participants in Group 1 were previously vaccinated at 12 to 18 months of age with a single dose of JE-CV vaccine and were to receive a booster dose of JE-CV vaccine on Day 0. This group was not randomized. JE vaccine naïve control children were randomized to receive one single dose of JE-CV on Day 0 (Group 2) or a varicella vaccination on Day 0 (Group 3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: JE-CV Vaccine Booster (Experimental): Participants previously vaccinated with JE-CV vaccine will receive a booster dose of JE-CV vaccine on Day 0.
  Interventions: Biological: JE-CV Vaccine
- Group 2: JE-CV Vaccine First Dose (Experimental): JE-CV vaccine naïve participants will receive a single dose of JE-CV vaccine on Day 0.
  Interventions: Biological: JE-CV Vaccine
- Group 3: Varicella Vaccine (Active Comparator): JE-CV vaccine naïve participants will receive one dose of Varicella vaccine on Day 0.
  Interventions: Biological: Varicella Vaccine

INTERVENTIONS:
Biological: JE-CV Vaccine — 0.5 mL (single dose), Subcutaneous
  Other Names: IMOJEV
  Arms: Group 1: JE-CV Vaccine Booster; Group 2: JE-CV Vaccine First Dose
Biological: Varicella Vaccine — 0.5 mL (single dose), Subcutaneous
  Other Names: OKAVAX®
  Arms: Group 3: Varicella Vaccine

SUMMARY:
The aim of the study is to investigate the memory immune response and the yearly persistence of the immunity against Japanese Encephalitis (JE) after vaccination with Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in participants previously vaccinated with JE-CV vaccine.

Objectives:

* To describe JE immune status before and after JE-CV vaccination in subjects previously vaccinated with JE-CV vaccine
* To describe the immune status before and after JE-CV vaccination in JE-naïve control subjects.
* To describe the safety (in terms of solicited and unsolicited adverse events) of a single dose of JE-CV vaccine up to 6 months after the last vaccination.
* To describe all related serious adverse events (SAEs) and related deaths from 6 months to 5 years after vaccination in JE-CV-primed subjects.

DETAILED DESCRIPTION:
Study participants who are previously immunized with JE-CV vaccine will receive a booster dose of the JE-CV vaccine and will be followed up for 5 years for immunogenicity.

The control (JE-CV naïve) participants will receive either one dose of JE-CV vaccine or one dose of varicella vaccine.

All participants will be monitored for safety for 6 month post-vaccination.

ELIGIBILITY:
An individual had to fulfill all of the following criteria in order to be eligible for trial enrollment:

All Participants

* Aged 36 to 42 months on the day of inclusion
* Provision of Informed Consent Form signed by at least one parent or other legally acceptable representative
* Participant and parent/legally acceptable representative or guardian able to attend all scheduled visits and to comply with all trial procedures
* In good general health, based on medical history and physical examination

For JE-CV vaccine primed group only

* Participant who was vaccinated with JE-CV in JEC02 trial (NCT00735644)

An individual fulfilling any of the following criteria was excluded from trial enrollment:

All Participants

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the Day 0 - Month 6 period and for Group 1 up to 5 years for any flavivirus vaccine trial
* Receipt of any vaccine* in the 4 weeks preceding the trial vaccination, except for pandemic influenza vaccination, which may be received at least 2 weeks before study vaccines
* Planned receipt of any vaccine* in the 4 weeks following the trial vaccination, except for pandemic influenza vaccine. In the event of local or national immunization program with a pandemic influenza vaccine, participants who receive a pandemic influenza vaccine at any time during the trial will not be withdrawn from the trial.
* Planned receipt of any JE vaccine during the course of the trial
* Administration of any anti-viral within 2 months preceding the trial vaccination and up to 4 weeks following the trial vaccination
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, as reported by the parent/legally acceptable representative
* History of central nervous system disorder or disease, including seizures and febrile seizures
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Chronic illness or any underlying illness (such as cardiovascular, kidney, liver or hematological disease or development abnormalities) that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion

  * Except in case of national immunization days with oral polio vaccine

For JE-CV primed participants only

* Receipt of any JE vaccine other than JE-CV during JEC02 trial(NCT00735644) and since the end of JEC02 trial

For JE-CV naïve participants only

* Previous vaccination against flavivirus disease including JE
* History of flavivirus infection either based on clinical suspicion or laboratory proven
* Previous vaccination against varicella
* Previous vaccination with JE-CV in JEC02 study
* History of varicella, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity or anaphylactic/anaphylactoid reaction to neomycin.
* Known history of thrombocytopenia or idiopathic thrombocytopenic purpura

Temporary Contraindications:

A prospective participant was not to be included in the study until the following conditions and/or symptoms had resolved:

1. Receipt of oral or injected antibiotic therapy within 72 hours prior to the first blood draw (for Groups 1 and 2)
2. Febrile illness (temperature ≥38.0°C [≥100.4°F]) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination (for all participants)

The Investigator was to postpone vaccination until the situation/condition resolved. Vaccination could be postponed within the timeframe for vaccination indicated in the protocol trial flowchart.

Ages: 36 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2010-08-25 (Actual); Primary Completion 2010-10-29 (Actual); Study Completion 2015-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Capeding MR, Alberto ER, Bouckenooghe A, Laot TM, Chansinghakul D, Monfredo C, Machabert T, Feroldi E. Five-Year Antibody Persistence Following a Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) Booster in JE-CV-Primed Children in the Philippines. J Infect Dis. 2018 Jan 30;217(4):567-571. doi: 10.1093/infdis/jix601. PMID 29325161
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 25 August 2010 to 12 October 2015 at 3 clinic sites in the Philippines.
Pre-assignment Details: A total of 454 participants who met all inclusion criteria and no exclusion criteria were enrolled in Group 1 or randomized to Group 2 or Group 3 on Day 0. All except 4 participants in Group 1 were vaccinated as planned (345 participants in Group 1, 46 participants in Group 2, and 59 participants in Group 3).
Groups:
- JE-CV Vaccine Booster: Participants previously received a single dose of JE-CV in the JEC02 trial and also received a booster dose of JE-CV in the current trial.
- JE-CV Vaccine First Dose: JE vaccine naïve control participants received a single dose of JE-CV on Day 0 (Immunogenicity Control group).
- Varicella Vaccine Group: JE vaccine naïve control participants received a varicella vaccination (Okavax®) on Day 0 (Safety Control group).
Period: Overall Study
Arm/Group | JE-CV Vaccine Booster | JE-CV Vaccine First Dose | Varicella Vaccine Group
Started | 349 | 46 | 59
Completed | 344 | 46 | 59
Not Completed | 5 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JE-CV Vaccine Booster | JE-CV Vaccine First Dose | Varicella Vaccine Group | Total
Number analyzed (Participants) | 345 | 46 | 59 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 345 | 46 | 59 | 450
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 39.6 (1.71) | 39.3 (1.99) | 39.3 (2.09) | 39.5 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 25 | 29 | 226
  Male | 173 | 21 | 30 | 224
Region of Enrollment [Number; unit: Participants]
  Philippines | 345 | 46 | 59 | 450

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With JE Seroprotection Before and Following a Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a 50% plaque reduction neutralization test (PRNT50). Seroprotection status for antibody levels against JE virus before (on Day 0) and after JE-CV vaccination (Day 7 and Day 28) was defined as neutralizing antibody titer ≥ 10 (1/dilution).
Time Frame: Day 0 (pre-vaccination) and Day 7 and Day 28 post-vaccination
Population: Seroprotection against JE-CV vaccine was assessed in the Per Protocol Analysis Set. Data for Varicella Vaccine Group were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Number; unit: Percentage of participants
Groups:
- JE-CV Booster: Participants previously received a single dose of JE-CV in the JEC02 trial and also received a booster dose of JE-CV in the current trial.
- JE-CV First Dose: JE naïve control participants received a single dose of JE-CV on Day 0 (Immunogenicity Control group).
Arm/Group | JE-CV Booster | JE-CV First Dose
Number analyzed (Participants) | 340 | 39
Percentage of participants
  Day 0 (pre-vaccination) | 80.3 | 0
  Day 7 post-vaccination | 96.2 | 15.4
  Day 28 post-vaccination | 100.0 | 89.7

2. Primary Outcome: Percentage of Participants With JE Seroconversion Following a Dose of Live Attenuated JE-CV Vaccine
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay. Seroconversion was defined as participants with a pre-vaccination titer <10 (1/dilution) and post-vaccination titer ≥10 (1/dilution, or participants with pre vaccination titer ≥10 (1/dilution) and a ≥4-fold increase from pre- to post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 7 and Day 28 post-vaccination
Population: Seroconversion was assessed in the Per Protocol Analysis Set. Data for Varicella Vaccine Group were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | JE-CV Booster | JE-CV First Dose
Number analyzed (Participants) | 340 | 39
Percentage of participants
  Day 7 post-vaccination | 66.8 | 15.4
  Day 28 post-vaccination | 95.3 | 89.7

3. Primary Outcome: Summary of Geometric Mean Titers of JE Virus Antibodies Following a Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) and Day 7 and Day 28 post-vaccination
Population: Geometric mean titers of JE virus antibodies were assessed in the Per Protocol Analysis Set. Data for Varicella Vaccine Group were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | JE-CV Booster | JE-CV First Dose
Number analyzed (Participants) | 340 | 39
Titers (1/dilution)
  Day 0 (pre-vaccination) | 39.4 [33.7 to 46.0] | 5.00 [5.00 to 5.00]
  Day 7 post-vaccination | 231 [191 to 279] | 6.41 [5.11 to 8.05]
  Day 28 post-vaccination | 2242 [1913 to 2628] | 178 [99.7 to 318]

4. Primary Outcome: Summary of Geometric Mean Titer Ratios of JE Virus Antibodies Following a Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) and Day 7 and Day 28 post-vaccination
Population: Geometric mean titer ratios of JE virus antibodies were assessed in the Per Protocol Analysis Set. Data for Varicella Vaccine Group were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios (1/dilution)
Groups:
- JE-CV Booster: Participants previously received a single dose of JE-CV Vaccine in the JEC02 trial and also received a booster dose of JE-CV in the current trial.
Arm/Group | JE-CV Booster | JE-CV First Dose
Number analyzed (Participants) | 340 | 39
Titer ratios (1/dilution)
  Day 7 post-vaccination | 5.87 [5.06 to 6.80] | 1.28 [1.02 to 1.61]
  Day 28 post-vaccination | 57.0 [47.8 to 67.9] | 35.6 [19.9 to 63.6]

5. Primary Outcome: Summary of Serological Flavivirus Status at Baseline of Participants Vaccinated With a Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay. Flavivirus positive was defined as titers against JE virus ≥10 (1/dilution) or titers against at least 1 dengue serotype ≥10 (1/dilution). Flavivirus negative was defined as titers against JE virus <10 (1/dilution) and titers against the 4 dengue serotypes <10 (1/dilution).
Time Frame: Day 0 (pre-vaccination)
Population: Serological flavivirus status at baseline was assessed in the Full Analysis Set. Data for Varicella Vaccine Group were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Number; unit: Number of participants
Arm/Group | JE-CV Booster | JE-CV First Dose
Number analyzed (Participants) | 345 | 46
Number of participants
  Any JE-CV and/or dengue virus; Flavivirus positive | 289 | 14
  Any JE-CV and/or dengue virus; Flavivirus negative | 56 | 32
  JE-CV virus strain | 277 | 7
  Any dengue serotype | 121 | 11
  Dengue serotype 1 | 116 | 11
  Dengue serotype 2 | 102 | 11
  Dengue serotype 3 | 96 | 9
  Dengue serotype 4 | 108 | 9

6. Primary Outcome: Percentage of Participants With JE Seroprotection Before and Up to 5 Years Following a Booster Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay. Seroprotection status for antibody levels against JE virus before (on Day 0) and after JE-CV vaccination (Days 7 and 28 and Years 1, 2, 3, 4, and 5) was defined as neutralizing antibody titer ≥ 10 (1/dilution).
Time Frame: Day 0 (pre-vaccination) and Days 7 and 28, and Year 1, 2, 3, 4, and 5 post-vaccination
Population: Seroprotection was assessed in the Full Analysis Set. Data for JE-CV Vaccine First Dose and Varicella Vaccine Groups were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | JE-CV Booster
Number analyzed (Participants) | 345
Percentage of participants
  Day 0 (pre-vaccination) | 80.3
  Day 7 post-vaccination | 96.2
  Day 28 post-vaccination: number analyzed (Participants) | 344
  Day 28 post-vaccination | 100.0
  Year 1 post-vaccination: number analyzed (Participants) | 339
  Year 1 post-vaccination | 99.4
  Year 2 post-vaccination: number analyzed (Participants) | 340
  Year 2 post-vaccination | 98.8
  Year 3 post-vaccination: number analyzed (Participants) | 338
  Year 3 post-vaccination | 99.1
  Year 4 post-vaccination: number analyzed (Participants) | 335
  Year 4 post-vaccination | 98.2
  Year 5 post-vaccination: number analyzed (Participants) | 336
  Year 5 post-vaccination | 98.2

7. Primary Outcome: Summary of Geometric Mean Titer of JE Virus Antibodies Before and Up to 5 Years Following a Booster Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) and Days 7 and 28 and Year 1, 2, 3, 4, and 5 post-vaccination
Population: Geometric mean titers of JE virus antibodies were assessed in the Full Analysis Set. Data for JE-CV Vaccine First Dose and Varicella Vaccine Groups were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | JE-CV Booster
Number analyzed (Participants) | 345
Titers (1/dilution)
  Day 0 (pre-vaccination) | 39.3 [33.7 to 45.8]
  Day 7 post-vaccination | 233 [193 to 281]
  Day 28 post-vaccination: number analyzed (Participants) | 344
  Day 28 post-vaccination | 2259 [1930 to 2645]
  Year 1 post-vaccination: number analyzed (Participants) | 339
  Year 1 post-vaccination | 596 [502 to 708]
  Year 2 post-vaccination: number analyzed (Participants) | 340
  Year 2 post-vaccination | 368 [313 to 432]
  Year 3 post-vaccination: number analyzed (Participants) | 338
  Year 3 post-vaccination | 301 [257 to 352]
  Year 4 post-vaccination: number analyzed (Participants) | 335
  Year 4 post-vaccination | 249 [215 to 289]
  Year 5 post-vaccination: number analyzed (Participants) | 336
  Year 5 post-vaccination | 161 [141 to 184]

8. Primary Outcome: Summary of Geometric Mean Titer Ratios of JE Virus Antibodies Up to 5 Years Following a Booster Dose of Live Attenuated JE-CV
Description: The presence of JE virus neutralizing antibodies was measured using a PRNT50 assay.
Time Frame: Year 1, 2, 3, 4, and 5 post-vaccination
Population: Geometric mean titer ratios of JE virus antibodies were assessed in the Full Analysis Set. Data for JE-CV Vaccine First Dose and Varicella Vaccine Groups were not analyzed for this outcome measure as pre-specified in the study protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios (1/dilution)
Arm/Group | JE-CV Booster
Number analyzed (Participants) | 345
Titer ratios (1/dilution)
  Year 2/Year 1: number analyzed (Participants) | 339
  Year 2/Year 1 | 0.615 [0.539 to 0.701]
  Year 3/Year 2: number analyzed (Participants) | 338
  Year 3/Year 2 | 0.821 [0.734 to 0.919]
  Year 4/Year 3: number analyzed (Participants) | 335
  Year 4/Year 3 | 0.827 [0.746 to 0.916]
  Year 5/Year 4: number analyzed (Participants) | 335
  Year 5/Year 4 | 0.646 [0.584 to 0.715]

9. Primary Outcome: Number of Participants With Solicited Injection-Site Reactions and Systemic Reactions Following a Dose of Live Attenuated JE-CV or Varicella Vaccine
Description: Injection-site reactions: Pain, Erythema, and Swelling. Systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 Injection-site reactions: Pain, Incapacitating, unable to perform usual activities. Erythema and Swelling, ≥5 cm. Grade 3 Systemic reactions: Fever, 39.0°C; Headache, Malaise, and Myalgia, Significant; prevents daily activities.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Groups:
- Varicella Vaccine Group: JE naïve control participants received a varicella vaccination (Okavax®) on Day 0 (Safety Control group).
Arm/Group | JE-CV Booster | JE-CV First Dose | Varicella Vaccine Group
Number analyzed (Participants) | 345 | 46 | 59
Participants
  Injection-site Pain: number analyzed (Participants) | 344 | 46 | 59
  Injection-site Pain | 73 | 13 | 12
  Grade 3 Injection-site Pain: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Injection-site Pain | 0 | 0 | 0
  Injection-site Erythema: number analyzed (Participants) | 344 | 46 | 59
  Injection-site Erythema | 29 | 1 | 4
  Grade 3 Injection-site Erythema: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Injection-site Erythema | 0 | 0 | 0
  Injection-site Swelling: number analyzed (Participants) | 344 | 46 | 59
  Injection-site Swelling | 19 | 0 | 1
  Grade 3 Injection-site Swelling: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Injection-site Swelling | 0 | 0 | 0
  Fever: number analyzed (Participants) | 344 | 46 | 59
  Fever | 49 | 1 | 9
  Grade 3 Fever: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Fever | 6 | 1 | 0
  Headache: number analyzed (Participants) | 344 | 46 | 59
  Headache | 41 | 5 | 8
  Grade 3 Headache: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Headache | 2 | 0 | 0
  Malaise: number analyzed (Participants) | 344 | 46 | 59
  Malaise | 49 | 6 | 6
  Grade 3 Malaise: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Malaise | 2 | 0 | 0
  Myalgia: number analyzed (Participants) | 344 | 46 | 59
  Myalgia | 19 | 2 | 2
  Grade 3 Myalgia: number analyzed (Participants) | 344 | 46 | 59
  Grade 3 Myalgia | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up Day 14 post-vaccination for solicited AEs, up to Day 28 post-vaccination for unsolicited AEs, and up to 5 years post-vaccination for SAEs.
Groups:
- JE-CV Vaccine Booster: Participants previously received a single dose of JE-CV Vaccine in the JEC02 trial and also received a booster dose of JE-CV in the current trial.
Arm/Group | JE-CV Vaccine Booster | JE-CV Vaccine First Dose | Varicella Vaccine Group
All-Cause Mortality (participants affected / at risk) | 0/345 | 0/46 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/345 | 0/46 | 0/59
Other Adverse Events (participants affected / at risk) | 73/345 | 13/46 | 12/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-CV Vaccine Booster (N=345) | JE-CV Vaccine First Dose (N=46) | Varicella Vaccine Group (N=59)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-CV Vaccine Booster (N=345) | JE-CV Vaccine First Dose (N=46) | Varicella Vaccine Group (N=59)
Rhinitis (Infections and infestations) | 12 (12) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 37 (41) | 3 (4) | 6 (6)
Injection site Pain (General disorders) | 73 (73) | 13 (13) | 12 (12)
Injection site Erythema (General disorders) | 29 (29) | 1 (1) | 4 (4)
Injection site Swelling (General disorders) | 19 (19) | 0 (0) | 1 (1)
Fever (General disorders) | 49 (49) | 1 (1) | 9 (9)
Headache (Nervous system disorders) | 41 (41) | 5 (5) | 8 (8)
Malaise (General disorders) | 49 (49) | 6 (6) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications